CLINICAL TRIAL: NCT04292561
Title: Effects of Different Sevoflurane Concentrations on Intraoperative EEG and Postoperative Delirium in Elderly Patients
Brief Title: Intraoperative EEG Monitoring and Postoperative Delirium in Elderly Patients With Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201912
Record Dates: First submitted 2020-01-08; First posted 2020-03-03 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Delirium; Sevoflurane; Electroencephalogram
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- light general anesthesia (Experimental): During anesthesia maintenance, patients were received with low concentration sevoflurane to maintain a target of 0.8 MAC.
  Interventions: Drug: Low MAC
- deep general anesthesia (Experimental): During anesthesia maintenance, patients were received with high concentration sevoflurane to maintain a target of 1.0 MAC.
  Interventions: Drug: High MAC

INTERVENTIONS:
Drug: Low MAC — To maintain a target of sevoflurane inhalation concentration 0.8 MAC.
  Arms: light general anesthesia
Drug: High MAC — To maintain a target of sevoflurane inhalation concentration 1.0 MAC.
  Arms: deep general anesthesia

SUMMARY:
Delirium is an acute onset of attentional and cognitive impairment. BIS guided anesthesia can reduce the incidence of postoperative delirium. Long term electroencephalogram (EEG) suppression during operation is related to postoperative delirium. The latest research shows that the anesthesia depth guided by EEG does not reduce the incidence of postoperative delirium. The purpose of this study was to explore the relationship between anesthesia exposure with different minimum alveolar concentration(MAC) and postoperative delirium(POD), and to observe the characteristics of EEG.

DETAILED DESCRIPTION:
More and more studies have focused on the relationship between EEG inhibition and postoperative delirium in general anesthesia. At present, there are two kinds of commonly processed quantitative EEG monitoring to evaluate the depth of anesthesia, one is bispectral index (BIS) and the other is patient state index (PSI). The relationship between intraoperative anesthetic exposure and postoperative delirium is unclear, or whether potential patient characteristics increase the risk of EEG suppression and postoperative delirium.

Gastrointestinal surgery can lead to long-term changes in colonic flora, which can remotely regulate brain function through the gut brain axis. We speculated that the abnormal composition of intestinal flora before abdominal operation might be the influencing factor of POD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastrointestinal diseases
* Patients were aged 60 to 90 years
* American Society of Anesthesiologists (ASA) risk classification II-IV
* Patients were scheduled to undergo elective major abdominal operation(with a anticipated time of 2-6 h)

Exclusion Criteria:

* Preoperative dementia or cognitive impairment
* Mental instability or mental illness
* Patients with any factors affecting cognitive assessment, such as language, vision and hearing impairment
* Any cerebrovascular accident occurred within 3 months, such as stroke etc
* Previous history of delirium
* Known hypersensitivity to sevoflurane or history of malignant hyperthermia
* Abuse of narcotic sedative and analgesic drugs
* Those who have reoperation within 7 days after operation

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Incidence of POD | The 1st day after the surgery
  Incidence of POD after surgery
Incidence of POD | The 2nd day after the surgery
  Incidence of POD after surgery
Incidence of POD | The 3rd day after the surgery
  Incidence of POD after surgery
Incidence of POD | The 5th day after the surgery
  Incidence of POD after surgery
Incidence of POD | The 7th day after the surgery
  Incidence of POD after surgery

SECONDARY OUTCOMES:
EEG burst inhibition | During surgery
  Frequency of EEG burst inhibition
EEG burst inhibition | During surgery
  Duration of EEG burst inhibition
Incidence of adverse events | 30-day after surgery
  Incidence of adverse events after surgery
length of stay | From 1st day after the surgery to 2 weeks
  length of stay after surgery
30-day mortality | 30-day after surgery
  30-day mortality after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xuesheng Liu, MD.PHD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Background] Chaput AJ, Bryson GL. Postoperative delirium: risk factors and management: continuing professional development. Can J Anaesth. 2012 Mar;59(3):304-20. doi: 10.1007/s12630-011-9658-4. Epub 2012 Feb 4. English, French. PMID 22311257
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Wildes TS, Mickle AM, Ben Abdallah A, Maybrier HR, Oberhaus J, Budelier TP, Kronzer A, McKinnon SL, Park D, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Goswami S, Jordan K, Lin N, Fritz BA, Stevens TW, Jacobsohn E, Schmitt EM, Inouye SK, Stark S, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):473-483. doi: 10.1001/jama.2018.22005. PMID 30721296
- [Background] Ridaura V, Belkaid Y. Gut microbiota: the link to your second brain. Cell. 2015 Apr 9;161(2):193-4. doi: 10.1016/j.cell.2015.03.033. PMID 25860600